CLINICAL TRIAL: NCT06428162
Title: an Observational Study for the Prevalence of Pharmacovigilance Practices Between Healthcare Providers in North African Nation
Brief Title: An Evaluation of Healthcare Providers' Adherence to Pharmacovigilance Practices in an African Community
Status: Completed | Type: Observational
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, associate professor of pharamcy practices, faculaty of pharmacy, Deraya University, Deraya University
Other Study IDs: 2024 PV
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Drug Reaction; Drug Hypersensitivity; Drug Abuse; Drug Interaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Drug Hypersensitivity; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionner — three sections questioner including: demographics, reported cases, unreported cases

SUMMARY:
Egypt's several regions-rural, mixed, and urban-were given pre-designed surveys pertaining to drug adverse events and the role of pharmacovigilance in detection and reporting. The three sections of the survey were dedicated to studying health care professionals' knowledge concerning pharmacovigilance concepts and practices, as well as demographics and people reported or not reported. The survey also asked more questions regarding adverse occurrences that were reported.

ELIGIBILITY:
Inclusion Criteria:

* all health care providers are invited to share in the study
* minimum experience required is one year in health carrier.
* accept sharing in the study

Exclusion Criteria:

* health care providers who refuse to complete all data required in the survey.
* fresh experience or participants who left health carrier

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all health care providers that deals with drugs and medications as pharmacists, physicians, Dentists, nurses and medical reps are invited to share in this survey as a hard template. study included 300 subject in different disciplines at the period at 3 months. complete survey composed of 3 sections included previous reported ADVEs
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
reported adverse drug reactions | 3 months
  collect recent adverse drug reaction reports

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Minya, Egypt